CLINICAL TRIAL: NCT05624671
Title: Is Elective Caesarean Sections for Predicting Post-spinal Hypotension Role of Overactive Bladder?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Professor Doctor, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: B.30.2ATA.0.01.00/
Record Dates: First submitted 2022-09-23; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: 18-45 Range of Age; Cesarean Section; Primigravid
Keywords: cesarean section; spinal-epidural; overactive bladder; post-spinal hypotension
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IS THERE ANY ROLE OF OVERACTIVE BLADDER IN POSTSPINAL HYPOTENSION IN ELECTIVE CAESAREAN SECTIONS? (Other): According to our institution protocol, intravenous (iv) hydration will not be given as preload and afterload and vasopressor infusion will not be initiated before spinal anesthesia. After the skin is prepared sterile and local infiltration with 2% lidocaine is done, from L3-L4 OR L4-L5 range on midline with the 16 gauge Tuohy needle and the loss of resistance technique epidural space is identified and then 26 gauge pencil point needle is passed trough the Touhy and the dura will be drilled. After the cerebrospinal fluid (CSF) is seen the fluid containing 5mg isobaric bupivacaine and 15µg fentanyl will be given in 30 seconds to patients. After the spinal needle is removed, the epidural catheter is placed 3-5 cm in the epidural space through Tuohy, and after the catheter is fixated, the patients will be placed in the supine position by placing a height under their right hip with a 15 ° angle.
  Interventions: Other: bupivacaine,fentanyl

INTERVENTIONS:
Other: bupivacaine,fentanyl — According to our institution protocol, intravenous (iv) hydration will not be given as preload and afterload and vasopressor infusion will not be initiated before spinal anesthesia. After the skin is prepared sterile and local infiltration with 2% lidocaine is done, from L3-L4 OR L4-L5 range on midline with the 16 gauge Tuohy needle and the loss of resistance technique epidural space is identified and then 26 gauge pencil point needle is passed trough the Touhy and the dura will be drilled. After the cerebrospinal fluid (CSF) is seen the fluid containing 5mg isobaric bupivacaine and 15µg fentanyl will be given in 30 seconds to patients. After the spinal needle is removed, the epidural catheter is placed 3-5 cm in the epidural space through Tuohy, and after the catheter is fixated, the patients will be placed in the supine position by placing a height under their right hip with a 15 ° angle.

SUMMARY:
It is to predict postspinal hypotension that may develop in patients diagnosed with overactive bladder who will undergo elective cesarean section under spinal-epidural anesthesia.

DETAILED DESCRIPTION:
INTRODUCTION

Spinal anesthesia is the most preferred standard anesthesia technique in caesarean sections. After a C-section, hypotension develops in approximately 70% of pregnant women and 33% of nonpregnant women and this situation is generally more severe and sudden in pregnant women. Aortocaval compression and low basal vasomotor tone caused by the Gravid Uterus and sympathetic blockade associated with spinal anesthesia contribute to this sudden onset and deep hypotension. Serious post-spinal hypotension that is not properly treated can increase the risks of maternal and fetal complications. It is important to identify patients at high risk of developing hypotension. Because it will enable us to manage the process more proactively.

Many predictive methods such as thoracic electrical bioimpedance, heart rate (HR) variability, pupillary light reflex analysis, and perfusion index (PI) were used to predict the onset of hypotension. In some studies, it has been shown that hypotension may develop with disruption of the balance between sympathetic and parasympathetic nervous systems in the autonomic nervous system.

The bladder is an organ in which the sympathetic and parasympathetic system works in coordination. For a normal micturition, the balance between the sympathetic and parasympathetic systems should not be disturbed. Overactive bladder (OAB) is a syndrome that includes symptoms such as sudden and severe urination, urge to urinate suddenly, incontinence before reaching the toilet, and frequent urination (≥8 per day). Overactive bladder can be diagnosed based on subjective symptoms instead of urodynamic tests. In our country, the rate is 20% for males, 35.7% for females and 29.3% for both sexes. The main problem here is the balance disturbed between the sympathetic and parasympathetic systems.

Our primary goal in the study is to predict post-spinal hypotension that may develop in patients with a diagnosis of the overactive bladder who will undergo elective cesarean under combined spinal epidural anesthesia.

MATERIALS AND METHODS

These randomized triple-blind prospective studies will be performed on the primiparous pregnant woman in ASA I-II, 2nd and 3rd trimester, who will undergo an elective caesarean under combined spinal epidural anesthesia after obtaining informed written consent from patients and the ethics office of Medicine Research Hospital of Atatürk University. Exclusion criteria: ≤18 or ≥45 years of age, emergency obstetric surgery, pregnancy-induced hypertension, significant systemic disease, multiple pregnancy, fetal or placental abnormality, hypersensitivity or allergy history to drugs to be used in the study, morbid obesity (BMI≥40), autonomic neuropathy, diabetes, patients with contraindications to neuraxial anesthesia, multigravida, urinary tract infection, and Cre≥1.2, who are unable or unwilling to participate in the study will be excluded. Patients diagnosed with OAB will be classified as Group I and other patients will be classified as Group II. Patients will be randomly assigned to Group I and Group II. For this, a random number table will be used.

ANESTHESIC MANAGEMENT

After patients have transferred to the operation room, an intravenous (iv) access is obtained with an applicator size of 20, and routine monitorization consisting of electrocardiogram (ECG), peripheral oxygen saturation (SpO2), and non-invasive blood pressure is performed. While the patient is in the supine and lateral tilt positions, blood pressure and heart rate will be measured 2 times consecutively and the average of these values will be recorded as a baseline value. From the beginning of spinal anesthesia to the end of surgery Isolyte S will be infused at room temperature with 10 mL/kg / h speed to patients. According to our institutional protocol, intravenous (iv) hydration will not be given as preload, and afterload and vasopressor infusion will not be initiated before spinal anesthesia. After the skin is prepared sterile and local infiltration with 2% lidocaine is done, from L3-L4 OR L4-L5 range on midline with the 16 gauge Tuohy needle, and the loss of resistance technique epidural space is identified and then 26 gauge pencil point needle is passed trough the Touhy and the dura will be drilled. After the cerebrospinal fluid (CSF) is seen the fluid containing 5mg isobaric bupivacaine and 15µg fentanyl will be given in 30 seconds to patients. After the spinal needle is removed, the epidural catheter is placed 3-5 cm in the epidural space through Tuohy, and after the catheter is fixated, the patients will be placed in the supine position by placing a height under their right hip with a 15 ° angle. Blankets will be used to maintain the body temperature of patients and all fluids used during surgery will be delivered at 24 ° C. Oxygen will be given to patients at 4l / min with a face mask throughout the operation.

OVERACTIVE BLADDER DIAGNOSIS

The presence of OAB for each patient in the primipara who applied in the second and third trimesters will be determined using the Turkish version of OAB-V8, which consists of eight questions that can be graded on a 6-point scale ranging from 0 to 5; 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit), 4 (a great deal) and 5 (a very great deal). The lowest total score will be 0, the highest total score will be 40, and those with a higher score than 11 will be evaluated in favor of OAB. With the OAB-V8 form, a non-invasive uroflowmetry test will be applied to pregnant women, and tower-like diagram will be interpreted in favor of OAB.

STUDY PROTOCOLS

After the spinal anesthesia has been performed in the following first 10 minutes blood pressure and heart rate will be measured in every minute after the first 10 minutes will be measured in every 2.5 minutes until the baby is born. Hypotension will be defined as symptom complaints compatible with hypotension (ex: paleness, dizziness, shortness of breath, nausea or vomiting) without the systolic blood pressure falling below 20% or systolic blood pressure below 20% of the basal value. If hypotension occurs, it will be treated with ephedrine until blood pressure reaches baseline (initial dose 10 mg, intravenously) and rapid colloid or crystalloid infusion. If hypotension persists or recurs, vasopressor treatment will be repeated every 1 minute. Bradycardia will be described as having a heart rate of 50 beats/min and will be treated with 1mg iv atropine. The spinal anesthesia will be considered as unsuccessful if the sensorial block level has not reached the T6 level before surgery or felt pain during skin incision. In this case, 10 ml of 15 ml 2% lidocaine + 2 ml bicarbonate + 2 ml fentanyl + 1ml 1/200000 adrenaline solution will be given via epidural catheter and the patient will be excluded from the study. However, if pain felt again, will switch to general anesthesia. Post-spinal hypotension will be recorded from the onset of spinal anesthesia to the birth of the fetus. After the completion of the C-section, the time until the skin incision, uterine incision and time of birth, and the height, weight, BMI, and trimester of patients will be recorded. After the birth of the fetus, the study will be terminated and the total dose of ephedrine, adrenaline, and atropine used, as well as the amount of crystalloid, and colloid administered, and blood loss will be recorded. The study was triple-blind because the researchers who detected, recorded, and treated post-spinal hypotension did not know the results obtained from urological measurements and did not know about the groups analyzed by the statistician.

STATISTICAL ANALYSIS

Power analysis : Patients diagnosed with OAB are 15% more likely to develop hypotension than patients who do not receive this diagnosis. In order for a difference of 15% to be statistically significant, it was calculated by the PAS statistics program, which requires a total of 142 patients to be included in the study, where 71 patients should be in each group at a 95% confidence level at 80% power.

The analyzes were done with IBM SPSS 20 statistical analysis program.

Data were presented as mean, standard deviation, median, minimum, maximum, percentage, and number. The normal distribution of continuous variables was evaluated with the Shapiro Wilk-W test when the sample size was <50 and the Kolmogorov-Smirnov test when it was> 50.

In the comparisons between two independent groups, the Independent Samples t test was used when the normal distribution condition was met and the Mann Whitney u test was used when it was not provided.

In 2x2 comparisons between categorical variables, the expected value (> 5) was made using the Pearson Chi-square test, the expected value (3-5) was made using the chi-square yacht test and the expected value (<3) using Fisher's Exact test.

The statistical significance level was taken as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Primigravid
* Elective cesarean sections

Exclusion Criteria:

* ≤18 age
* ≥45 age
* Emergency surgery
* Pregnancy-induced hypertension,
* Significant systemic disease,
* Multiple pregnancy,
* Fetal or placental abnormality,
* History of hypersensitivity or allergy to drugs to be used in the study,
* Morbidly obese (BMI≥40),
* Patients for whom neuraxial anesthesia is contraindicated,
* Unable or unwilling to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 143 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Is Elective Caesarean Sections for Predicting Post-spinal Hypotension (reduction of systolic blood pressure(mmHg) after spinal anesthesia) Role of Overactive Bladder? | Intraoperative period
  It is to predict postspinal hypotension (systolic blood pressure below 20% of the basal value) that may develop in patients diagnosed with overactive bladder who will undergo elective cesarean section under spinal-epidural anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞENUR DOSTBİL, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided